CLINICAL TRIAL: NCT00670722
Title: Observational Study on Evaluation of Glycaemic Control in Patients Using a Modern Insulin - NovoRapid® (Insulin Aspart), NovoMix® 30 (Biphasic Insulin Aspart 30) or Levemir® (Insulin Detemir) for Treatment of Type 2 Diabetes Mellitus
Brief Title: Observational Study on Blood Glucose Control in Patients With Diabetes Using Modern Insulin
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3517
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin Detemir; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A
  Interventions: Drug: insulin aspart
- B
  Interventions: Drug: insulin detemir
- C
  Interventions: Drug: biphasic insulin aspart 30
- D
  Interventions: Drug: insulin aspart; Drug: insulin detemir

INTERVENTIONS:
Drug: insulin aspart — Intervention at the discretion of the physician
  Other Names: NovoRapid®
  Groups: A; D
Drug: insulin detemir — Intervention at the discretion of the physician
  Groups: B; D
Drug: biphasic insulin aspart 30 — Intervention at the discretion of the physician
  Groups: C

SUMMARY:
This study is conducted in Europe. An observational study evaluating the blood glucose control in patients using a modern insulin: NovoRapid®, NovoMix® 30 or Levemir® for treatment of Type 2 diabetes mellitus in Czech Republic.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Current treatment with human soluble insulin, insulin NPH or premixed human insulin
* The selection of the subjects will be at the discretion of the individual physician

Exclusion Criteria:

* Current treatment with insulin aspart, insulin detemir or biphasic insulin aspart 30
* Previous enrolment in this study
* Hypersensitivity to insulin aspart, insulin detemir or biphasic insulin aspart 30 or to any of the excipients.
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within next 6 months and considered to be treated by biphasic insulin aspart 30 or insulin detemir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
HbA1c after switch from human insulin to modern insulin treatment | After 24 weeks

SECONDARY OUTCOMES:
Percentage of subjects to reach HbA1c below 7.0% and = 6.5% at approximately 12 weeks and 24 weeks of treatment | After 12 and 24 weeks
Postprandial glycaemic control as measured by PPG | After 12 and 24 weeks
Glucose variability as measured by FPG | After 12 and 24 weeks
Insulin dose and number of injections | After 12 and 24 weeks
Body weight | After 12 and 24 weeks
Number of hypoglycaemic events | During treatment
Number of adverse drug reactions (ADR) | After 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Prague, Czechia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com